CLINICAL TRIAL: NCT03012490
Title: Efficacy, Safety and Cost of Comprehensive Versus Standard Remote Monitoring of Patients With Cardiac Resynchronization Therapy
Brief Title: Efficacy, Safety and Cost of Remote Monitoring of Patients With Cardiac Resynchronization Therapy
Acronym: ECOST-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Biotronik France (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016_03; 2016-A00873-48 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-12-19; First posted 2017-01-06 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure; Cardiac Resynchronization Therapy
Keywords: Remote monitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard remote monitoring (Active Comparator): Remote monitoring of CRT-P and CRT-D is activated. The physician will only receive the notifications related to technical events and ventricular arrhythmias. Therapy will be added or changed in response to these notifications and/or the symptoms and signs observed during ambulatory visits.
  Interventions: Other: CRT-P or CRT-D standard remote monitoring
- Comprehensive remote monitoring (Experimental): Remote monitoring of CRT-P and CRT-D is activated, as well as remote assessment of symptoms and signs. In addition to notifications related to technical events and ventricular arrhythmias, the physician will receive notifications related to heart failure parameters, atrial arrhythmias, and patient's symptoms and signs. Therapy will be added or changed in response to these notifications, and/or to the symptoms and signs observed during ambulatory visits.
  Interventions: Other: CRT-P or CRT-D standard remote monitoring; Other: CRT-P or CRT-D full remote monitoring; Other: Symptoms and signs remote monitoring

INTERVENTIONS:
Other: CRT-P or CRT-D standard remote monitoring — standard for the control group: remote monitoring of ventricular rhythm disorders and technical parameters of the implanted system
Other: CRT-P or CRT-D full remote monitoring — Full follow-up for the Active group: remote monitoring of ventricular rhythm disorders and technical parameters of the implanted system + supraventricular rhythm disorders, parameters related to heart failure, including symptoms and clinical signs of the patient
  Arms: Comprehensive remote monitoring
Other: Symptoms and signs remote monitoring — symptoms and clinical signs of the patient
  Arms: Comprehensive remote monitoring

SUMMARY:
The primary objective is to determine whether comprehensive remote follow-up in HF patients with CRT will reduce the combined endpoint of all-cause mortality or worsening heart failure hospitalizations, whichever comes first, when compared to basic remote monitoring, over a 27-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient more than 18 years old, newly implanted, in accordance to the latest European guidelines, with a CRT-P or CRT-D device (upgrading is tolerated but no device replacement), with Home-Monitoring® activated
* Patient willing and able to comply with the protocol and who has provided written informed consent

Exclusion Criteria:

* Lead model under advisory
* Non-functional lead except particular case of non-functional or deactivated right atrial lead due to atrial fibrillation
* Known drug or alcohol abuse
* Pregnant woman or woman who plan to become pregnant during the trial (the data will be collected by querying the patient without a pregnancy test is required)
* Participation (ongoing or planned during the trial) in another interventional clinical study, and/or another remote monitoring and/or follow-up concept, unless authorized by the Executive Committee
* Participation (ongoing or planned during the trial) in an investigational HF program (e.g. PRADO, PIMPS, OSICAT, CARDIAUVERGNE)
* Estimated life-expectancy, regardless of the cardiovascular condition, <1year
* Patient under- or planned for - ventricular assistance
* Patient not living in Metropolitan France and/or not geographically stable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
composite criteria including death from any cause and hospitalization for worsening HF | during the 27 months follow-up

SECONDARY OUTCOMES:
Costs including hospital costs for unplanned cardiovascular hospitalizations, medical charges for ambulatory follow-up of CRT devices and transportation related costs | 27 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Guedon-Moreau, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Institut coeur poumon, CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Klein C, Kouakam C, Lazarus A, de Groote P, Bauters C, Marijon E, Mouquet F, Degand B, Guyomar Y, Mansourati J, Leclercq C, Guedon-Moreau L; ECOST-CRT study Investigators. Comprehensive vs. standard remote monitoring of cardiac resynchronization devices in heart failure patients: results of the ECOST-CRT study. Europace. 2024 Oct 3;26(10):euae233. doi: 10.1093/europace/euae233. PMID 39400005